CLINICAL TRIAL: NCT01412996
Title: Single Access Laparoscopic Cholecystectomy
Brief Title: Quality of Life Measures After Single Access Vs Conventional Laparoscopic Cholecystectomy: Prospective Randomized Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MOHAMED ABDELLATIF, ASS. PROF., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Single access chOLECYSTECTOMY
Record Dates: First submitted 2011-08-04; First posted 2011-08-09 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Evidence of Cholecystectomy
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single ACCESS cholecystectomy (Active Comparator): single ACCESS laparoscopic cholecystectomy
  Interventions: Procedure: surgery
- traditional (Active Comparator): conventional laparoscopic cholecystectomy
  Interventions: Other: SURGERY

INTERVENTIONS:
Procedure: surgery — single ACCESS laparoscopic cholecystectomy
  Other Names: SALC; GROUP I
  Arms: single ACCESS cholecystectomy
Other: SURGERY — CONVENTIONAL LAPAROSCOPIC CGOLECYSTECTOMY
  Other Names: CLC; GROUP II
  Arms: traditional

SUMMARY:
This study aimed to compare the short term outcomes between SALC and conventional laparoscopic cholecystectomy (CLC).

DETAILED DESCRIPTION:
In a prospective study, two hundred fifty patients with symptomatic gall bladder stone were randomized to SALC or conventional laparoscopic cholecystectomy (CLC) (125 in each group). The primary endpoint of this study was to assess the total outcomes of quality of life using EuroQoL EQ-5D questionnaire. The secondary endpoints were postoperative pain, analgesia requirement and duration, operative time, perioperative complications, estimated blood loss, hospital stay, cosmoses outcomes and number of days required to return to normal activities.

ELIGIBILITY:
Inclusion Criteria:

* GALL BLADDER STONES

Exclusion Criteria:

* ACUTE CHOLECYSTITIS
* PREVIOUS LAPAROTOMY
* ASA ABOVE 3

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
QUALITY OF LIFE | PREOPERATIVEELY, after 1 WEEK, 1 and 6 months postoperative
  Quality of life was the primary endpoint of this study assessed by EuroQoL EQ-5D 9 questionnaire preoperatively, 1 week, 1 and 6 months after surgery. The EQ-5D is a validated questionnaire which consists of 2 pages: the EQ-5D descriptive system and EQ visual analogue scale (EQ VAS). The WQ-5D-descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.

SECONDARY OUTCOMES:
operative time | 2 hours
  (defined as the interval between the initial skin incision and skin closure)
postoperative pain | 5 days
  using verbal analogue scale (VAS) from 0 to 10 (0 = no pain, 10 = severe pain)
days to return to normal activity (RTNA) | 10 days
  patients were contacted by phone every day until they are able to return to their normal daily works
COSMOSIS OUTCOMES | 1 AND 6 MONTHS
  cosmetic outcomes 1 and 6 months after surgery using Patient and Observer Scar Assessment Scale (POSAS)(10), it comprises two distinct series of Visual Analogue Scale (VAS) instruments: one is self-assessed by the patient and one by an independent doctor, ranging from 1 (poor) to 10 (excellent)
ANALGESIC REQUIRMENT | POSTOPERATIVE PERIOD
  NOMBERS OF ANALGESIC TABLETS AND NO. OF DAYS ANALGESIA NEEDED

CONTACTS AND LOCATIONS:
Overall Officials: RAMADAN ELLITHY, MD, Study Chair — Mansoura University
Locations (1):
- Mohamed Abdellatif, Al Mansurah, Egypt